CLINICAL TRIAL: NCT07367412
Title: Effect of Zinc Supplementation on Occurrence of Infections in Older Medical Patients (ZOOM) - a Cluster Randomized Controlled Trial (ZOOM OUT).
Brief Title: Zinc Supplementation and Infections in Older Medical Patients
Acronym: ZOOM OUT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Independent Research Fund Denmark (Industry); The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Cecilia Margareta Lund, Associate Professor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZOOM OUT
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Older Adults (65 Years and Older); Medical Patients in the Emergency Department
Keywords: Older adults; Infections; Days alive and out of hospital; Zinc supplementation
MeSH Terms: conditions — Infections | interventions — Zinc; Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: The study is a cluster randomized controlled trial. Patients ≥ 65 years referred to the Medical Emergency Department at Herlev Hospital, and meet the inclusion criteria, will be randomized to participate in the study.
  Randomization In EPIC (Sundhedsplatformen) a generic module has been developed that facilitate cluster-level randomization directly in the system. In this study, clusters of time, will be used to randomly assign groups of patients to intervention with zinc supplementation (intervention n = 1000), recommendation of zinc supplementation (recommendation n = 3000), or usual care (control n = 4000). An automatic pop-up in EPIC (Sundhedsplatformen) will occur when a doctor opens the patients electronic medical chart. The randomization will occur based on unequal time windows with the same ratio of hours (8:6:2 hours) to ensure the anticipated segregation of 4:3:1. The time windows will be shifting an agreed number of minutes every day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Active Comparator): The intervention group will consist of 1000 patients who following discharge from the hospital will have daily zinc supplements prescribed and provided free of charge which will be sent to their home for a year.
  Interventions: Dietary Supplement: Zinc (zinc sulphate)
- Recommendation group (Experimental): The recommendation group will consist of 3000 patients who will have zinc supplements recommended and prescribed. However, zinc supplements will not be provided free of charge.
  Interventions: Dietary Supplement: Zinc (zinc sulphate)
- Control group (No Intervention): The control group will consist of 4000 patients who will receive usual care

INTERVENTIONS:
Dietary Supplement: Zinc (zinc sulphate) — 22 mg zinc sulphate tablets taken once daily for 12 months
  Arms: Intervention; Recommendation group

SUMMARY:
The goal of this clinical trial is to learn about the effect of zinc supplementation once daily for 12 months in older acute medical patients. The main question it aims to answer is:

• Can daily zinc supplementation for 12 months increase Days Alive and Out of Hospital (DAOH)? Researchers will compare zinc supplementation to a control group, a group who do not receive zinc supplementation, to see if zinc supplementation can increase Days Alive and Out of Hospital, reduce antibiotic use, readmissions and mortality.

Participants will take 22 mg zinc supplementation once daily for 12 months or not.

The researchers will draw data on readmissions, antibiotic use and mortality during the 12 months follow-up period.

DETAILED DESCRIPTION:
1. Study purpose Older adults are at increased risk of micronutrient deficiencies, including zinc, due to sparse food intake. Zinc deficiency is known to increase the susceptibility to infections, further exacerbating the vulnerability of older adults to health complications. Infections are common among older adults and are a leading causes of acute hospital admissions and readmissions.

   The hypothesis is that zinc supplementation for older acutely admitted medical patients can increase Days Alive and Out of Hospital regardless of baseline plasma zinc level

   Objectives:

   Primary objective: To test in older acute medical patients if zinc supplementation once daily for 12 months can increase Days Alive and Out of Hospital.

   Secondary objectives: To evaluate if zinc supplementation once daily can reduce antibiotic use, readmissions and mortality during the 12 months follow-up period.
2. Short background A large proportion of older adults are malnourished, which can lead to increased morbidity, mortality, prolonged hospitalization and reduced quality of life (QoL). With malnutrition the patient lacks vitamins and minerals, including zinc, which is essential for older adults. Early detection and treatment of malnutrition has been shown to be beneficial for patients, including reducing length of stay in the hospital. The older adults are at increased risk of zinc deficiency, with less than half of the free-living older adults having a sufficient zinc intake. Zinc is essential for immune function and acute deficiency weakens both innate and adaptive immunity, increasing susceptibility to infections. The effects of zinc supplementation on infections are conflicting, some studies do not find an effect of zinc supplementation in patients with infections, while other studies of healthy or institutionalized older adults, found that zinc supplementation significantly reduce the incidence of infections, antibiotic use and prevention of symptomatic COVID-19. Despite previous findings, the effect of zinc supplementation has not been studied in older acutely admitted medical patients on a large scale.
3. Method This study is a cluster randomized controlled trail. A total of 8000 patients will be included and divided into three groups. Patients ≥ 65 years, who come to the Medical Emergency Department at Herlev Hospital, and who meet the inclusion criteria, will be offered participations in the study. An automatic pop-up in the patient medical record will appear in blocks of time and will randomly assign patients to intervention with zinc supplementation (intervention n = 1000), recommendation of zinc supplementation (recommendation n = 3000) or control (n = 4000), regardless of plasma zinc levels at admission. The treating doctor will assess if the patient is eligible and include the patient to the study.

   Measurements and collection of clinical data Date on readmissions and mortality will be collected from the electronic medical chart EPIC (Sundhedsplatformen). Data on prescribed antibiotics will be drawn from the Danish National Prescription Register. Antibiotic prescriptions within 15 days, will be considered as a single treatment, as described in a previous study.

   Research plan Project "ZOOM" will be included in a PhD programme. Inclusion is expected to start in February 2026. The inclusion period is anticipated to span 12 months, followed by a 12-month intervention period. Consequently, the intervention period ends in January 2028.

   Assessment of compliance To minimize waste of zinc supplements, patients in the intervention group will be contacted every 3 months, to assess further need of zinc supply, which will reflect the adherence of intervention.
4. Statistical consideration

   1. Power calculation No available data exists to estimate the primary endpoint of Days Alive and Out of Hospital 12 months after acute hospitalization of older medical patients. However, a previous study that investigated this for patients with non-STEMI found a mean (SD) of 273 (123) days. Assuming that zinc supplementation can increase days alive and out of the hospital with 3% (8 days), we estimated a sample size of approximately 7422 patients (3712 in each arm), with an estimated power of 80%, 2-sided α-level of 0.05. Due to an estimated rate of loss to follow-up of approximately 10 %, we aim to enroll 8000 patients in the study. We plan to randomize participants into three groups: intervention, recommendation and control. However, the intervention and recommendation group will be considered as a single group for analysis. We plan to include patients during a 1-year study period. About 16.900 older patients (≥ 65 years) are hospitalized to the Medical Emergency Department, Herlev Hospital every year.
   2. Plan for statistical analysis of data Categorical variables will be compared using Chi-square test where appropriate; otherwise, Fisher's exact test will be used. Descriptive analyses of continuous variables will be per-formed using the Wilcoxon rank sum test. Binary outcomes will be analyzed by logistic re-gression and presented as odds ratios (ORs) and 95% confidence intervals (Cis). Overall sur-vival (OS) will be analyzed by the Kaplan Meier estimator; hazard ratios (HRs) and 95% CIs will be estimated by Cox proportional hazards regression. The primary endpoint (Days Alive and Out of Hospital) will be compared as a continuous variable between the two groups us-ing the analysis of variance test.
5. Risks, adverse events and disadvantages

   a. Safety measures that minimize pain, discomfort, fear, and other risks All patients will receive standard treatment during and after hospitalization. The intervention group receives one capsule of 22 mg zinc sulfate once daily for 12 months. This dose is based on an assessment of achieving efficacy in reducing infections, improve immune function, while also being safe, with no serious adverse effects. The dose is far from the toxic zinc level of 1-2 grams per day, with no risk of serious adverse effects and below the U.S. Food and Drug Administration (40 mg/day). Adverse events of the zinc in doses around 22 mg daily are mild and most often consist of gastrointestinal symptoms (nausea, upset stomach, dizziness) and dry mouth. In a recent Cochrane review, it was not possible to distinguish between adverse events cause by zinc supplementation and events caused by the cold itself (e.g. headache).

   Chronic zinc toxicity leads to copper deficiency with bone marrow (granulocytopenia, sideroblastic anemia, myelodysplastic syndrome) and neurologic effects (ascending, sen-sorimotor polyneuropathy syndrome). Copper deficiency is the most serious adverse event of long-term zinc overdose. The daily zinc dose at 45 mg has previously been shown to be safe in a healthy cohort of older adults; by not reducing plasma-copper and at the same time the zinc supplementation significantly reduced the number of infections. Zinc is not considered being carcinogenic in general. A 30-year follow-up study showed that low zinc intake < 9mg/day may increase the risk of prostate cancer, whereas extremely high doses of > 75 mg/day and long-term supplementation could increase the risk of aggressive prostate cancer.
6. Information from patient records We will not use medical records without consent.

   Specific information will be collected for implementation of the trial:
   * Age, to evaluate if certain age-groups could benefit more from zinc supplementation than others.
   * Results of routine blood parameters (CRP, neutrophils, leucocytes, platelets, hemoglobin, electrolytes, creatinine, eGFR, liver enzymes, lipids, HbA1c)
   * Weight, height
   * Demographic data
   * Results of routinely assess Clinical Frailty Scale
   * Disease history and the number of ICD-10 discharge diagnoses 5 years prior to admission, to assess comorbidity.
   * Number of medications and type of medication at admission, to evaluate polypharmacy
   * Length of hospitalization
   * Readmission, cause and number of days admitted within 6 and 12 months
   * Antibiotic use within 6 and 12 months
   * Date of death and cause or day of follow-up if alive at 12 months after inclusion
7. Processing of personal data in the project Data will be handled in accordance with The Data Protection Regulation and the Data Protection Act. The study is approved by the Danish National Medical Research Ethics Committee (VMK) and the Danish Data Protection Agency, before inclusion of patients. Data will be stored up to 5 years after end of study.

   Patient discontinuation Discontinuation may occur if the participant withdraws consent to participate in the study and/or withdraws consent for the use of their data. If a participant withdraws their consent, they will not be included in the study and their data will not be stored or analyzed. Information related to withdrawal will be obtained through "Sundhedsplatformen". The participant will be informed that they can withdrawal their consent at any time. Participants will receive a digital letter, two weeks after discharge, describing their participations in the study and informing them of their right to withdraw consent.
8. Finances The study has received funding from the "Independent Research Fund Denmark", "Herlev and Gentofte Hospital Internal PhD Fellowship Funds", "Clinical Academic Groups", and "Novo Nordic Foundation". The investigators have no financial ties to the sponsor, or any other interests related to the trial.
9. Recruitment of participants and informed consent

   a. Recruitment of participants This is a cluster randomized trial, in which each cluster consists of time. The treating doctor will assess if the patient is eligible (none of the exclusion criteria are present) and then include the patient.
10. Publication and sharing data Results from the study, both negative, inconclusive, and positive, will be published in rele-vant peer-reviewed international scientific journals The investigators will be co-authors on all publications according to Vancouver guidelines. The project will be reported according to CONSORT guidelines and registered at www.clinicaltrials.gov before initiation.
11. Patient insurance All participants are secured via the Danish Patient Compensation.

ELIGIBILITY:
Inclusion Criteria:

* All medical patients aged ≥ 65 years assessed at the Medical Emergency Department, Herlev Hospital

Exclusion Criteria:

* Self-supplementing with zinc at time of assessment (> 10 mg zinc/day)
* Terminal illness (life expectancy < 6 months, estimated by Clinical Frailty Scale ≥8)
* Patients receiving parenteral nutrition (partial or complete)
* Patients treated with hemodialysis or peritoneal dialysis
* Patients know with known severe dementia
* Patients who do not understand Danish and patients with temporary civil person registration numbers (CPR)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Days Alive and Out of Hospital | During the 12 months follow-up period
  To evaluate the differences between the groups in Days Alive and Out of Hospital. The endpoints will include date of death, date of hospitalization, and number of days hospitalized during the 12 months follow-up period in the three groups

SECONDARY OUTCOMES:
Antibiotic use | During the 12 months follow-up period
  Number of episodes with use of antibiotic
Hospital admissions | During the 12 months follow-up period
  Number of hospital episodes of any cause
Readmission due to cardiovascular disease | During the 12 months follow-up period
  Number of readmissions due to cardiovascular disease
Readmissions due to infections | During the 12 months follow-up period
  Number of readmissions due to infections
Mortality | During the 12 months follow-up period
  Number of deaths

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Copenhagen University Hospital - Herlev and Gentofte, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be avilable from January 2029 to 2034 and
Access Criteria: Will be available from the corresponding author upon reasonable request and only after approval has been granted by an ethics committee.

REFERENCES:
- [Background] Hopewell S, Chan AW, Collins GS, Hrobjartsson A, Moher D, Schulz KF, Tunn R, Aggarwal R, Berkwits M, Berlin JA, Bhandari N, Butcher NJ, Campbell MK, Chidebe RCW, Elbourne D, Farmer A, Fergusson DA, Golub RM, Goodman SN, Hoffmann TC, Ioannidis JPA, Kahan BC, Knowles RL, Lamb SE, Lewis S, Loder E, Offringa M, Ravaud P, Richards DP, Rockhold FW, Schriger DL, Siegfried NL, Staniszewska S, Taylor RS, Thabane L, Torgerson D, Vohra S, White IR, Boutron I. CONSORT 2025 statement: updated guideline for reporting randomised trials. BMJ. 2025 Apr 14;389:e081123. doi: 10.1136/bmj-2024-081123. PMID 40228833
- [Background] European Parliament C of the EU. EU regulation No 536/2014 of the European parliaments and of the council of 16th of April 2014 on clinical trials on pharmaceutical products for human use article 30 (informed consent in cluster trials). http://data.europa.eu/eli/reg/2014/536/2022-12-05 2014
- [Background] Zhang Y, Song M, Mucci LA, Giovannucci EL. Zinc supplement use and risk of aggressive prostate cancer: a 30-year follow-up study. Eur J Epidemiol. 2022 Dec;37(12):1251-1260. doi: 10.1007/s10654-022-00922-0. Epub 2022 Nov 3. PMID 36326979
- [Background] Porea TJ, Belmont JW, Mahoney DH Jr. Zinc-induced anemia and neutropenia in an adolescent. J Pediatr. 2000 May;136(5):688-90. doi: 10.1067/mpd.2000.103355. PMID 10802505
- [Background] Nault D, Machingo TA, Shipper AG, Antiporta DA, Hamel C, Nourouzpour S, Konstantinidis M, Phillips E, Lipski EA, Wieland LS. Zinc for prevention and treatment of the common cold. Cochrane Database Syst Rev. 2024 May 9;5(5):CD014914. doi: 10.1002/14651858.CD014914.pub2. PMID 38719213
- [Background] Silk R, LeFante C. Safety of zinc gluconate glycine (Cold-Eeze) in a geriatric population: a randomized, placebo-controlled, double-blind trial. Am J Ther. 2005 Nov-Dec;12(6):612-7. doi: 10.1097/01.mjt.0000179115.04316.18. PMID 16280656
- [Background] Institute of Medicine (US) Panel on Micronutrients. Dietary Reference Intakes for Vitamin A, Vitamin K, Arsenic, Boron, Chromium, Copper, Iodine, Iron, Manganese, Molybdenum, Nickel, Silicon, Vanadium, and Zinc. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222310/ PMID 25057538
- [Background] Plum LM, Rink L, Haase H. The essential toxin: impact of zinc on human health. Int J Environ Res Public Health. 2010 Apr;7(4):1342-65. doi: 10.3390/ijerph7041342. Epub 2010 Mar 26. PMID 20617034
- [Background] Bao B, Prasad AS, Beck FW, Fitzgerald JT, Snell D, Bao GW, Singh T, Cardozo LJ. Zinc decreases C-reactive protein, lipid peroxidation, and inflammatory cytokines in elderly subjects: a potential implication of zinc as an atheroprotective agent. Am J Clin Nutr. 2010 Jun;91(6):1634-41. doi: 10.3945/ajcn.2009.28836. Epub 2010 Apr 28. PMID 20427734
- [Background] Intorre F, Polito A, Andriollo-Sanchez M, Azzini E, Raguzzini A, Toti E, Zaccaria M, Catasta G, Meunier N, Ducros V, O'Connor JM, Coudray C, Roussel AM, Maiani G. Effect of zinc supplementation on vitamin status of middle-aged and older European adults: the ZENITH study. Eur J Clin Nutr. 2008 Oct;62(10):1215-23. doi: 10.1038/sj.ejcn.1602844. Epub 2007 Jul 11. PMID 17622255
- [Background] Duncan A, Morrison I, Bryson S. Iatrogenic copper deficiency: Risks and cautions with zinc prescribing. Br J Clin Pharmacol. 2023 Sep;89(9):2825-2829. doi: 10.1111/bcp.15749. Epub 2023 May 25. PMID 37070154
- [Background] Prasad AS. Essentiality and toxicity of zinc. Scand J Work Environ Health. 1993;19 Suppl 1:134-6. No abstract available. PMID 8159965
- [Background] Boukaiba N, Flament C, Acher S, Chappuis P, Piau A, Fusselier M, Dardenne M, Lemonnier D. A physiological amount of zinc supplementation: effects on nutritional, lipid, and thymic status in an elderly population. Am J Clin Nutr. 1993 Apr;57(4):566-72. doi: 10.1093/ajcn/57.4.566. PMID 8460613
- [Background] Girodon F, Galan P, Monget AL, Boutron-Ruault MC, Brunet-Lecomte P, Preziosi P, Arnaud J, Manuguerra JC, Herchberg S. Impact of trace elements and vitamin supplementation on immunity and infections in institutionalized elderly patients: a randomized controlled trial. MIN. VIT. AOX. geriatric network. Arch Intern Med. 1999 Apr 12;159(7):748-54. doi: 10.1001/archinte.159.7.748. PMID 10218756
- [Background] Sanchis J, Bueno H, Minana G, Guerrero C, Marti D, Martinez-Selles M, Dominguez-Perez L, Diez-Villanueva P, Barrabes JA, Marin F, Villa A, Sanmartin M, Llibre C, Sionis A, Carol A, Garcia-Blas S, Calvo E, Morales Gallardo MJ, Elizaga J, Gomez-Blazquez I, Alfonso F, Garcia Del Blanco B, Nunez J, Formiga F, Ariza-Sole A. Effect of Routine Invasive vs Conservative Strategy in Older Adults With Frailty and Non-ST-Segment Elevation Acute Myocardial Infarction: A Randomized Clinical Trial. JAMA Intern Med. 2023 May 1;183(5):407-415. doi: 10.1001/jamainternmed.2023.0047. PMID 36877502
- [Background] Bjork E, Aabenhus R, Larsen SP, Ryg J, Henriksen DP, Lundby C, Pottegard A. Use of antibiotics for urinary tract infections up to and after care home admission in Denmark: a nationwide study. Eur Geriatr Med. 2024 Jun;15(3):797-805. doi: 10.1007/s41999-024-00976-1. Epub 2024 May 2. PMID 38698277
- [Background] Gordon AM, Hardigan PC. A Case-Control Study for the Effectiveness of Oral Zinc in the Prevention and Mitigation of COVID-19. Front Med (Lausanne). 2021 Dec 13;8:756707. doi: 10.3389/fmed.2021.756707. eCollection 2021. PMID 34966750
- [Background] Girodon F, Lombard M, Galan P, Brunet-Lecomte P, Monget AL, Arnaud J, Preziosi P, Hercberg S. Effect of micronutrient supplementation on infection in institutionalized elderly subjects: a controlled trial. Ann Nutr Metab. 1997;41(2):98-107. doi: 10.1159/000177984. PMID 9267584
- [Background] Prasad AS, Beck FW, Bao B, Fitzgerald JT, Snell DC, Steinberg JD, Cardozo LJ. Zinc supplementation decreases incidence of infections in the elderly: effect of zinc on generation of cytokines and oxidative stress. Am J Clin Nutr. 2007 Mar;85(3):837-44. doi: 10.1093/ajcn/85.3.837. PMID 17344507
- [Background] Berti AD, Kale-Pradhan PB, Giuliano CA, Aprilliano BN, Miller CR, Alyashae BT, Bhargava A, Johnson LB. Clinical Outcomes of Zinc Supplementation Among COVID-19 Patients. Curr Drug Saf. 2022;17(4):366-369. doi: 10.2174/1574886317666220317115023. PMID 35301954
- [Background] Douglas RM, Miles HB, Moore BW, Ryan P, Pinnock CB. Failure of effervescent zinc acetate lozenges to alter the course of upper respiratory tract infections in Australian adults. Antimicrob Agents Chemother. 1987 Aug;31(8):1263-5. doi: 10.1128/AAC.31.8.1263. PMID 3307620
- [Background] Turner RB, Cetnarowski WE. Effect of treatment with zinc gluconate or zinc acetate on experimental and natural colds. Clin Infect Dis. 2000 Nov;31(5):1202-8. doi: 10.1086/317437. Epub 2000 Nov 6. PMID 11073753
- [Background] Bonaventura P, Benedetti G, Albarede F, Miossec P. Zinc and its role in immunity and inflammation. Autoimmun Rev. 2015 Apr;14(4):277-85. doi: 10.1016/j.autrev.2014.11.008. Epub 2014 Nov 24. PMID 25462582
- [Background] Prasad AS. Discovery of human zinc deficiency: its impact on human health and disease. Adv Nutr. 2013 Mar 1;4(2):176-90. doi: 10.3945/an.112.003210. PMID 23493534
- [Background] Berger MM, Shenkin A, Schweinlin A, Amrein K, Augsburger M, Biesalski HK, Bischoff SC, Casaer MP, Gundogan K, Lepp HL, de Man AME, Muscogiuri G, Pietka M, Pironi L, Rezzi S, Cuerda C. ESPEN micronutrient guideline. Clin Nutr. 2022 Jun;41(6):1357-1424. doi: 10.1016/j.clnu.2022.02.015. Epub 2022 Feb 26. PMID 35365361
- [Background] Mocchegiani E, Romeo J, Malavolta M, Costarelli L, Giacconi R, Diaz LE, Marcos A. Zinc: dietary intake and impact of supplementation on immune function in elderly. Age (Dordr). 2013 Jun;35(3):839-60. doi: 10.1007/s11357-011-9377-3. Epub 2012 Jan 6. PMID 22222917
- [Background] Maret W, Sandstead HH. Zinc requirements and the risks and benefits of zinc supplementation. J Trace Elem Med Biol. 2006;20(1):3-18. doi: 10.1016/j.jtemb.2006.01.006. Epub 2006 Feb 21. PMID 16632171
- [Background] Kruizenga HM, Van Tulder MW, Seidell JC, Thijs A, Ader HJ, Van Bokhorst-de van der Schueren MA. Effectiveness and cost-effectiveness of early screening and treatment of malnourished patients. Am J Clin Nutr. 2005 Nov;82(5):1082-9. doi: 10.1093/ajcn/82.5.1082. PMID 16280442
- [Background] Schulz MT, Rink L. Zinc deficiency as possible link between immunosenescence and age-related diseases. Immun Ageing. 2025 May 19;22(1):19. doi: 10.1186/s12979-025-00511-1. PMID 40390089
- [Background] Wapnir RA. Zinc deficiency, malnutrition and the gastrointestinal tract. J Nutr. 2000 May;130(5S Suppl):1388S-92S. doi: 10.1093/jn/130.5.1388S. PMID 10801949
- [Background] Agarwal E, Miller M, Yaxley A, Isenring E. Malnutrition in the elderly: a narrative review. Maturitas. 2013 Dec;76(4):296-302. doi: 10.1016/j.maturitas.2013.07.013. Epub 2013 Aug 2. PMID 23958435
- [Background] Marshall S, Bauer J, Isenring E. The consequences of malnutrition following discharge from rehabilitation to the community: a systematic review of current evidence in older adults. J Hum Nutr Diet. 2014 Apr;27(2):133-41. doi: 10.1111/jhn.12167. Epub 2013 Nov 30. PMID 24289811
- [Background] Andersen AL, Nielsen RL, Houlind MB, Tavenier J, Rasmussen LJH, Jorgensen LM, Treldal C, Beck AM, Pedersen MM, Andersen O, Petersen J. Risk of Malnutrition upon Admission and after Discharge in Acutely Admitted Older Medical Patients: A Prospective Observational Study. Nutrients. 2021 Aug 11;13(8):2757. doi: 10.3390/nu13082757. PMID 34444917
- [Background] Goto T, Yoshida K, Tsugawa Y, Camargo CA Jr, Hasegawa K. Infectious Disease-Related Emergency Department Visits of Elderly Adults in the United States, 2011-2012. J Am Geriatr Soc. 2016 Jan;64(1):31-6. doi: 10.1111/jgs.13836. Epub 2015 Dec 23. PMID 26696501
- [Background] Buurman BM, Hoogerduijn JG, de Haan RJ, Abu-Hanna A, Lagaay AM, Verhaar HJ, Schuurmans MJ, Levi M, de Rooij SE. Geriatric conditions in acutely hospitalized older patients: prevalence and one-year survival and functional decline. PLoS One. 2011;6(11):e26951. doi: 10.1371/journal.pone.0026951. Epub 2011 Nov 14. PMID 22110598